CLINICAL TRIAL: NCT06422546
Title: A Prospective, Multicenter, Non-interventional, Real-world Study to Characterize Changes in Molecular Markers After Three Weeks of Targeted Therapy With Oxitinib in Chinese Patients With Stage IV Metastatic or Recurrent Non-squamous EGFR-positive NSCLC
Brief Title: A Prospective, Multicenter, Non-interventional, Real-world Study to Characterize Changes in Molecular Markers After Three Weeks of Targeted Therapy With Oxitinib in EGFRm NSCLC
Acronym: pre-FLAME
Status: Recruiting | Type: Observational
Sponsor: Beijing Cancer Prevention & Treatment Society (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: pre-FLAME
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EGFR mutation in plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the characteristics of genetic variationmutations at baseline and 3 weeks after oxitinib treatment in EGFRm NSCLC

DETAILED DESCRIPTION:
Characteristics of EGFR gene mutation and efficacy of oxitinib treatment at baseline and after 3 weeks of treatment.To evaluate the mechanism of oxitinib treatment resistance and describe the characteristics of genetic variation associated with oxitinib treatment at baseline and 3 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old male or female
2. Stage IV metastatic or recurrent non-squamous NSCLC that is newly diagnosed, histologically proven and not suitable for radical surgery or radiotherapy (AJCC V8);
3. Without prior systemic antitumor therapy including EGFR-TKI or immunotherapy;
4. EGFR positive in blood or tissue tested in local laboratory;
5. Sufficient blood samples can be provided for molecular detection;
6. Signed informed consent forms are available.

Exclusion Criteria:

1. Patients were unable to collect plasma samples at baseline;
2. The EGFR mutant status of the patient's blood specimen at baseline has not been verified by the central laboratory;
3. The patient refused subsequent treatment with oxitinib; 4）The investigator determines that may affect the conduct of the clinical study and the judgement of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stage IV metastatic or recurrent non-squamous EGFR-positive NSCLC
Sampling Method: Probability Sample
Enrollment: 950 (Estimated)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
changes in EGFR gene mutations | baseline and 3 weeks after oxitinib treatment
  To characterize the changes in EGFR gene mutations at baseline and 3 weeks after oxitinib treatment

SECONDARY OUTCOMES:
Characteristics of EGFR gene mutation and efficacy of oxitinib treatment | baseline and 3 weeks after oxitinib treatment
  Characteristics of EGFR gene mutation and efficacy of oxitinib treatment at baseline and after 3 weeks of treatment

OTHER OUTCOMES:
describe the characteristics of genetic variation associated with oxitinib treatment | baseline and 3 weeks after oxitinib treatment
  To evaluate the mechanism of oxitinib treatment resistance and describe the characteristics of genetic variation associated with oxitinib treatment at baseline and 3 weeks after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Prevention society, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No